CLINICAL TRIAL: NCT06503588
Title: Ureteral Stent Exchange Abstention in Urinary Tract Infections: a Before-and-after Study to Assess Guidelines' Impact on Patients' Outcomes
Brief Title: Ureteral Stent Exchange Abstention in Urinary Tract Infections
Acronym: JJ-change-UTI
Status: Recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, LEFEVRE Benjamin, MD. PhD., Central Hospital, Nancy, France
Other Study IDs: 2022PI037
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Urinary Tract Infections; Urinary Catheterization
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Before guidelines: Patients treated for ureteral stent associated urinary tract infection in the University Hospital of Nancy from January 1, 2018 to May 31, 2020
- After guidelines: Patients treated for ureteral stent associated urinary tract infection in the University Hospital of Nancy from August 1, 2020 to December 31, 2022
  Interventions: Other: Guidelines promoting surgical abstention

INTERVENTIONS:
Other: Guidelines promoting surgical abstention — Guidelines promoting surgical abstention
  Groups: After guidelines

SUMMARY:
The Committee of Infectiology of the French Association of Urology (CIAFU) provided, for the first time in 2020, comprehensive guidelines for ureteral stent-associated urinary tract infections (USAUTI) prevention, diagnosis and treatment. Since evidence lacked in terms of appropriate treatment, guidelines could not support systematic change of US in case of USAUTI.

This study aims to evaluate whether "after guidelines group" patients treated for USAUTI had different occurrence of at least one relapse or recurrence than "before guidelines group".

ELIGIBILITY:
Inclusion Criteria:

* All patients with indwelling ureteral catheter
* AND confirmed or probable urinary tract infection

Exclusion Criteria:

* Patient's opposition
* History of ileal conduit urinary diversion
* Second or more urinary tract infection during the study period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Groups will be selected from patients attending University Hospital of Nancy meeting the eligibility criteria during the period of inclusion running from January 1, 2018 to May 31, 2020 and from August 1, 2020 to December 31, 2022
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Relapse OR recurrence of urinary tract infection | 1 year

SECONDARY OUTCOMES:
Nephro-urologic complication | 1 year
  Acute kidney injury ; hematuria ; pain ; stent migration or incrustation
Infectious complication | 1 year
  Sepsis or septic shock
In-hospital and 1-year mortality | 1 year
  all cause death
Resort to Watch or Reserve antibiotics | 1 year
  antibiotics' WHO classifcation

CONTACTS AND LOCATIONS:
Overall Officials: +33383154097 Lefevre, M.D. PhD, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- Nancy university hospital, Nancy, Lorraine, France

IPD SHARING:
Plan to Share IPD: No